CLINICAL TRIAL: NCT04748107
Title: Treatment of Severe Hypertension With Impendence Cardiography (ICG) Directed Therapy; a Randomized Controlled Trial
Brief Title: Treatment of Severe Hypertension With ICG Directed Therapy
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Too difficult to perform study procedures prior to giving blood pressure medication.
Sponsor: Marshall University (Other)
Responsible Party: Principal Investigator, Jesse Cottrell, Assistant Professor, Marshall University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1605500
Record Dates: First submitted 2020-11-02; First posted 2021-02-10 (Actual); Last update posted 2023-06-13 (Actual); Status verified 2023-06

CONDITIONS: Hypertension in Pregnancy
MeSH Terms: conditions — Hypertension, Pregnancy-Induced

STUDY DESIGN:
Intervention Model Description: Randomization to treatment of non treatment group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Provider preference: Control group (No Intervention): Provider will prescribe blood pressure medication based on his professional expertise.
- ICG directed therapy group (Experimental): ICG directed therapy will be used to determine which blood pressure medication is received.
  Interventions: Diagnostic Test: Impendence Cardiography

INTERVENTIONS:
Diagnostic Test: Impendence Cardiography — ICG is a noninvasive method of determining the amount of blood flow using the Non-Invasive Cardiac System - Cardiac Surveyor (NICaS) system, which provides an assessment of the cardiovascular system, respiratory system, and fluid retention.
  Arms: ICG directed therapy group

SUMMARY:
The purpose of the study is to compare the usefulness of Impedence Cardiography (ICG) directed therapy in treating severe range hypertension in pregnant women at term.

DETAILED DESCRIPTION:
Research Protocol

Study Design: Randomized Control Trial This is a randomized control trial comparing the usefulness of impedance cardiography (ICG) directed therapy in treating severe range hypertension (systolic BP >160 OR diastolic BP >110) in patients greater than 20 weeks gestation. All patients in the study will receive standard of care medication within the suggested timeframe by the American College of Obstetrics and Gynecology (ACOG). All patients will receive a hemodynamic assessment prior to receiving and after receiving medications. The treatment patients will receive either labetalol or nifedipine therapy for hypertension based on their hemodynamic parameters. The control group will receive medication based on provider preference (which is the usual plan of care).

Study Population:

Patients presenting to Labor and Delivery at Cabell Huntington Hospital being treated for severe range blood pressures. Consent will be obtained prior to randomization to standard care or ICG directed care. Patient age range will be from age 15 to approximately 45.

Schedule of Assessment:

An interval assessment will be performed after 20 patients have been assessed. The goal is for a total enrollment of 100 patients, 50 to the ICG directed treatment group and 50 to the control group.

Study Procedures:

If a patient presents to Labor and Delivery at Cabell Huntington Hospital and consents to the study, she will be randomized to either the ICG directed therapy group or provider preference group. Patients from each group will receive a non-invasive hemodynamic assessment via the NICaS system. The NICaS system uses impedance cardiography which provides a reliable assessment of cardiovascular, respiratory, and fluid parameters. The vasodilator nifedipine will be initiated for increased systemic vascular resistance. Elevated cardiac output will be treated with beta blockade via IV labetalol. ACOG recommends either of these medications as first line therapy for elevated blood pressure, and offers no guidance on which medication should be used first. All patients who are being treated will receive the standard of care treatment, however the ICG group will receive therapy based on their hemodynamic parameters.

Study Analysis The control group will be compared to the ICG directed treatment group.

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting to Labor and Delivery at Cabell Huntington Hospital being treated for severe range blood pressure after 20 weeks gestation. Patients will be English speaking and range in ages from 15-45 years old. Patient's will be consented prior to randomization.

Exclusion Criteria:

* Patients presenting to Labor and Delivery at Cabell Huntington Hospital with normal range blood pressures, or those with elevated blood pressures who do not consent to the study, patients <20 weeks gestation, or patients with eclampsia.

Ages: 15 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — Pregnant women
Enrollment: 0 (Actual)
Dates: Start 2021-04-25 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-06-01 (Actual)

PRIMARY OUTCOMES:
The systolic blood pressure | 1 year
  mmHg
The diastolic blood pressure | 1 year
  mmHg
mean arterial pressure | 1 year
  mmHg
heart rate | 1 year
  beats/minute
cardiac output (L/min) | 1 year
  liters per minute
systemic vascular resistance | 1 year
  dynes · sec/cm^-5

CONTACTS AND LOCATIONS:
Overall Officials: Jesse Cottrell, MD, Principal Investigator — Marshall University
Locations (1):
- Cabell Huntington Hospital, Huntington, West Virginia, United States

IPD SHARING:
Plan to Share IPD: No